CLINICAL TRIAL: NCT05668949
Title: Phase I/II Open Label Study Evaluating the Safety and Efficacy of Combining STAT3 Inhibition (TTI-101) With Anti-PD-1 Therapy (Pembrolizumab) in Patients With Recurrent or Metastatic (RM) Head and Neck Squamous Cell Carcinoma (HNSCC)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI requested
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Tvardi Therapeutics, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0625; NCI-2022-10803 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-12-20; First posted 2022-12-30 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — C188-9 compound; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Dose Escalation) (Experimental): Participants will be assigned to a study part based on when you join this study
  Interventions: Drug: TTI-101; Drug: Pembrolizumab
- Part 2 (Dose Expansion) (Experimental): Participants will be assigned to a study part based on when you join this study.
  Interventions: Drug: TTI-101; Drug: Pembrolizumab

INTERVENTIONS:
Drug: TTI-101 — Given by PO
Drug: Pembrolizumab — Given by IV (vein)
  Other Names: KEYTRUDA®

SUMMARY:
To review safety and efficacy of TTI-101 plus Pembrolizumab in patients the Recurrent and Metastatic head and Neck Squamous Cell Carcinoma.

DETAILED DESCRIPTION:
Primary Objectives:

* Objective (Phase I): Determine the phase II dose of TTI-101 when used in combination with pembrolizumab in solid tumor patients.
* Objective (Phase II): Determine the overall response rate (ORR) and progression free survival (PFS) of the combination evaluated according to RECIST criteria.

Secondary Objectives:

* Objective: Determine the overall survival in HNSCC patients treated with the combination.
* Objective: Determine the rate of immune-related severe adverse events (irSAEs) of the combination.
* Objective: Evaluate the safety of the combination in solid tumor patients. Secondary Endpoint: Overall SAEs, SAEs resulting in death, discontinuation, dose reduction or dose interruption, frequency, and time to onset and severity of AEs.

Exploratory Objectives:

--Objective: Determine the relationship between pharmacokinetics, pharmacodynamics, baseline and post-treatment immune and tumor biomarkers and clinical responses in patients treated with the combination.

ELIGIBILITY:
Inclusion Criteria:

Participant Inclusion Criteria

Participants are eligible to be included in the study only if all the following criteria apply:

Inclusion Criteria - phase II only

1. Histologically or cytologically confirmed diagnosis of HNSCC for which no standard curative therapy is available.
2. No prior treatment with an anti-PD-1 antibody (e.g. nivolumab, pembrolizumab, cemiplimab), as well as anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.
3. Appropriate for single agent pembrolizumab.

   1. Front line therapy for those whose tumors express PD L1 (CPS ≥1) OR
   2. Front line therapy for those who cannot tolerate chemotherapy per the judgement of the treating physician OR
   3. As second line or greater line of therapy.

Inclusion Criteria - phase I only

1. Histologically or cytologically confirmed diagnosis of an invasive solid tumor malignancy, for which no standard curative or life prolonging therapy is available OR
2. Meets all inclusion criteria above for the phase II study.

Inclusion Criteria - both safety and phase II

1. Male/female participants who are at least 18 years of age on the day of signing informed consent.
2. A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.
3. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
   2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 120 days after the last dose of study treatment.
4. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
5. Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
6. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 21 days prior to the first dose of study intervention.
7. Have adequate organ function as defined in the following table (Table 4). Specimens must be collected within 14 days prior to the start of study intervention.
8. Able to swallow TT1-101 capsules whole.

Exclusion Criteria:

Participant Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to initiation of treatment (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has received prior systemic anti-cancer therapy including investigational agents within 3 weeks prior to initiation of treatment.

   Participants must have recovered from all AEs due to previous therapies to ≤ Grade 1 or baseline with the following exceptions: Participants with ≤ Grade 2 neuropathy are eligible. Participants with endocrine-related AEs Grade ≤2 requiring treatment or hormone replacement are eligible.
3. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
4. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed or mRNA vaccines is allowed.
5. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 3 weeks prior to the first dose of study intervention.
6. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
7. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ that have undergone potentially curative therapy are not excluded.
8. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
9. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
11. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
12. Has an active infection requiring systemic therapy.
13. Human Immunodeficiency Virus (HIV)-infected (HIV1/2 antibody-positive) patients may participate IF they meet all the following eligibility requirements:

    1. They must be on an anti-retroviral regimen with evidence of at least two undetectable viral loads within the past 6 months on this same regimen; the most recent undetectable viral load must be within the past 12 weeks.
    2. They must have a CD4 count ≥250 cells/mcL over the past 6 months on this same antiretroviral regimen and must not have had a CD4 count <200 cells/ mcL over the past 2 years, unless it was deemed related to the cancer and/or chemotherapy-induced bone marrow suppression.
    3. For patients who have received chemotherapy in the past 6 months, a CD4 count <250 cells/mcL during chemotherapy is permitted as long as viral loads were undetectable during this same chemotherapy.
    4. They must have an undetectable viral load and a CD4 count ≥250 cells/mcL within 7 days of enrolment.
    5. They must not be currently receiving prophylactic therapy for an opportunistic infection and must not have had an opportunistic infection within the past 6 months.
14. Has a known active Hepatitis B (defined as Hepatitis B RNA detected) or known active Hepatitis C virus (defined as HCV RNA is detected) infection.
15. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
16. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
17. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
18. Has had an allogenic tissue/solid organ or bone marrow transplant.
19. Significantly impaired cardiac function such as unstable angina pectoris, congestive heart failure with New York Heart Association (NYHA) class III or IV, myocardial infarction within the last 12 months prior to trial entry; signs of pericardial effusion, serious arrhythmia (including QTc prolongation of >470 ms and/or pacemaker) or prior diagnosis of congenital long QT syndrome or left ventricular ejection fraction <50% on screening echocardiogram.
20. History of cerebral vascular accident or stroke within the previous 2 years.
21. Uncontrolled hypertension (>160/100mm Hg).
22. History of Grade 3 or 4 allergic reactions attributed to compounds of similar chemical or biologic composition as TTI-101 (hydroxyl-naphthalene sulfonamides).
23. Previous treatment of the current malignancy with a STAT inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09-23 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Faye Johnson, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org